CLINICAL TRIAL: NCT00750594
Title: Patent Foramen Ovale in Children With Migraine Headaches
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Primary Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 00026512
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Migraine Headaches
Keywords: Children; Migraine headaches
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This study will be the first to provide data about the relationship between PFO and migraine in children. By establishing the actual prevalence, we will better understand if PFO plays a role in the occurence of pediatric migraine and, thus, provide the incentive to perform additional studies evaluating whether PFO closure is an effective treatment option for pediatric migraine. For children with migraine headaches, discovering novel and effective treatments would be life altering.

DETAILED DESCRIPTION:
Specific Aim 1 Using contrast transthoracic echocardiography, compare the prevalence of a PFO in children with migraine headache with the established incidence of PFO published for the general population.

Specific Aim 2 Using contrast transcranial Doppler, examine the relationship between the degree of right to left atrial shunting with the presence or absence of aura in children with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to six years of age and less than 18 years of age.
* Diagnosis of migraine headache based on the International Headache Society Criteria.
* English speaking patients (and parent/guardians where appropriate).
* Signed informed consent/assent (as appropriate) given by patient, parent or legal guardian.

Exclusion Criteria:

* Inability to cooperate with imaging studies.
* Known congenital heart disease.
* Parent or guardian is unwilling to have their child undergo contrast echocardiography.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric neurology clinic
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The prevalence of PFO in children with migraine headaches | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rachel McCandless, MD, Principal Investigator — University of Utah; LuAnn Minich, MD, Study Chair — University of Utah; James Bale, MD, Study Chair — University of Utah
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Stewart WF, Lipton RB, Celentano DD, Reed ML. Prevalence of migraine headache in the United States. Relation to age, income, race, and other sociodemographic factors. JAMA. 1992 Jan 1;267(1):64-9. PMID 1727198
- [Result] Goadsby PJ, Lipton RB, Ferrari MD. Migraine--current understanding and treatment. N Engl J Med. 2002 Jan 24;346(4):257-70. doi: 10.1056/NEJMra010917. No abstract available. PMID 11807151
- [Result] Lauritzen M. Pathophysiology of the migraine aura. The spreading depression theory. Brain. 1994 Feb;117 ( Pt 1):199-210. doi: 10.1093/brain/117.1.199. PMID 7908596
- [Result] Olesen J, Larsen B, Lauritzen M. Focal hyperemia followed by spreading oligemia and impaired activation of rCBF in classic migraine. Ann Neurol. 1981 Apr;9(4):344-52. doi: 10.1002/ana.410090406. PMID 6784664
- [Result] Agmon Y, Khandheria BK, Meissner I, Gentile F, Sicks JD, O'Fallon WM, Whisnant JP, Wiebers DO, Seward JB. Comparison of frequency of patent foramen ovale by transesophageal echocardiography in patients with cerebral ischemic events versus in subjects in the general population. Am J Cardiol. 2001 Aug 1;88(3):330-2. doi: 10.1016/s0002-9149(01)01656-3. No abstract available. PMID 11472723
- [Result] Hagen PT, Scholz DG, Edwards WD. Incidence and size of patent foramen ovale during the first 10 decades of life: an autopsy study of 965 normal hearts. Mayo Clin Proc. 1984 Jan;59(1):17-20. doi: 10.1016/s0025-6196(12)60336-x. PMID 6694427
- [Result] Del Sette M, Angeli S, Leandri M, Ferriero G, Bruzzone GL, Finocchi C, Gandolfo C. Migraine with aura and right-to-left shunt on transcranial Doppler: a case-control study. Cerebrovasc Dis. 1998 Nov-Dec;8(6):327-30. doi: 10.1159/000015875. PMID 9774749
- [Result] Anzola GP, Magoni M, Guindani M, Rozzini L, Dalla Volta G. Potential source of cerebral embolism in migraine with aura: a transcranial Doppler study. Neurology. 1999 May 12;52(8):1622-5. doi: 10.1212/wnl.52.8.1622. PMID 10331688
- [Result] Domitrz I, Mieszkowski J, Kaminska A. Relationship between migraine and patent foramen ovale: a study of 121 patients with migraine. Headache. 2007 Oct;47(9):1311-8. doi: 10.1111/j.1526-4610.2006.00724.x. PMID 17927647
- [Result] Schwerzmann M, Nedeltchev K, Lagger F, Mattle HP, Windecker S, Meier B, Seiler C. Prevalence and size of directly detected patent foramen ovale in migraine with aura. Neurology. 2005 Nov 8;65(9):1415-8. doi: 10.1212/01.wnl.0000179800.73706.20. Epub 2005 Sep 7. PMID 16148260
- [Result] Dalla Volta G, Guindani M, Zavarise P, Griffini S, Pezzini A, Padovani A. Prevalence of patent foramen ovale in a large series of patients with migraine with aura, migraine without aura and cluster headache, and relationship with clinical phenotype. J Headache Pain. 2005 Sep;6(4):328-30. doi: 10.1007/s10194-005-0223-9. PMID 16362702
- [Result] Wilmshurst P,Dowson A,Muir K,Mullen M,Nightingale S. The prevalence and size of persistent foramen ovale in migraine patients: Preliminary results from the migraine intervention with STARFlex (R) technology (MIST) trial [abstract]. Circulation 2005; 112:3051.
- [Result] Post MC, Budts W. The relationship between migraine and right-to-left shunt: Fact or fiction? Chest. 2006 Sep;130(3):896-901. doi: 10.1378/chest.130.3.896. PMID 16963692
- [Result] Slavin L, Tobis JM, Rangarajan K, Dao C, Krivokapich J, Liebeskind DS. Five-year experience with percutaneous closure of patent foramen ovale. Am J Cardiol. 2007 May 1;99(9):1316-20. doi: 10.1016/j.amjcard.2006.12.054. Epub 2007 Mar 20. PMID 17478165
- [Result] Kimmelstiel C, Gange C, Thaler D. Is patent foramen ovale closure effective in reducing migraine symptoms? A controlled study. Catheter Cardiovasc Interv. 2007 Apr 1;69(5):740-6. doi: 10.1002/ccd.21025. PMID 17295330
- [Result] Schwerzmann M, Wiher S, Nedeltchev K, Mattle HP, Wahl A, Seiler C, Meier B, Windecker S. Percutaneous closure of patent foramen ovale reduces the frequency of migraine attacks. Neurology. 2004 Apr 27;62(8):1399-401. doi: 10.1212/01.wnl.0000120677.64217.a9. PMID 15111681
- [Result] Shammas NW, Dippel EJ, Harb G, Egts S, Jerin M, Stoakes P, Byrd J, Shammas GA, Sharis P. Interatrial septal defect closure for prevention of cerebrovascular accidents: impact on recurrence and frequency of migraine headaches. J Invasive Cardiol. 2007 Jun;19(6):257-60. PMID 17541126
- [Result] Anzola GP, Frisoni GB, Morandi E, Casilli F, Onorato E. Shunt-associated migraine responds favorably to atrial septal repair: a case-control study. Stroke. 2006 Feb;37(2):430-4. doi: 10.1161/01.STR.0000199082.07317.43. Epub 2005 Dec 22. PMID 16373630
- [Result] Thanigaraj S, Valika A, Zajarias A, Lasala JM, Perez JE. Comparison of transthoracic versus transesophageal echocardiography for detection of right-to-left atrial shunting using agitated saline contrast. Am J Cardiol. 2005 Oct 1;96(7):1007-10. doi: 10.1016/j.amjcard.2005.05.061. PMID 16188533